CLINICAL TRIAL: NCT02175290
Title: Machado-Joseph Disease in Israel: Clinical Phenotype and Genotype of a Jew Yemenite Subpopulation
Brief Title: Machado-Joseph Disease in Israel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC140006CTIL
Record Dates: First submitted 2014-06-22; First posted 2014-06-26 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2016-04

CONDITIONS: Spinocerebellar Ataxia 3
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinocerebellar Ataxia 3 Yemenite Jews patients

SUMMARY:
Machado-Joseph disease (MJD) or spinocerebellar ataxia type 3 (SCA-3) is the most common dominant ataxia. The genetic cause of this late-onset degenerative disorder is the expansion of a (CAG)n tract located in the exonic region of the ATXN3 gene. In 1994 the first case of MJD among the Yemenite Jewish subpopulation living in Israel was published. The puropse of this study is to describe the clinical phenotype and genotype of the Yemenite Jewish subpopulation with MJD living in Israel

ELIGIBILITY:
Inclusion Criteria:

* Spinocerebellar Ataxia 3 Yemenite Jews patients

Exclusion Criteria:

* All others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinocerebellar Ataxia 3 Yemenite Jews patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
clinical phenotype of SCA3 Yemenite Jews patients | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided